CLINICAL TRIAL: NCT06527313
Title: Investigation of the Effect of Movement Mobilization Concept on Quantitative Sensory Parameters, Pain, Muscle Activation Levels in Patients With Knee Osteoarthritis
Brief Title: Investigation of the Effect of Movement Mobilization Concept on Sensory, Pain, Muscle Activation in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Burcu Pamukcu, research assistant, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BI-1
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Osteo Arthritis Knee; Movement Disorders; Physical Disability; Knee Osteoarthritis
Keywords: osteoartritis; movement mobilization concept; mulligan; knee; taping
MeSH Terms: conditions — Movement Disorders; Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: . The study will be planned as a parallel research with 3 groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The research was designed as a double-blind randomized controlled study in which the participant and the evaluator were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Movement Mobilization Concept Group (Experimental): MWM and appropriate taping will be applied to the cases included in the Mulligan group, according to the Mulligan Concept, and home exercises will be given to the patient as recommended by the concept.
  Interventions: Behavioral: Movement Mobilization Concept, Exercise and Tape
- Sham Movement Mobilization Concept Group (Sham Comparator): The technique will be applied to cases in the sham group with only hand contact, without any slippage or rotation in any direction. Then, rigid taping will be applied without any tension or direction, and home exercises will be given.
  Interventions: Behavioral: Sham Movement Mobilization Concept, Exercise and Tape
- Control Group (Active Comparator): Subjects in the control group will be shown home exercises customized for knee osteoarthritis and asked to continue them.
  Interventions: Behavioral: Special Exercises

INTERVENTIONS:
Behavioral: Movement Mobilization Concept, Exercise and Tape — Mulligan Concept MWM Mulligan Taping Mulligan Self Home Workout
  Arms: Movement Mobilization Concept Group
Behavioral: Sham Movement Mobilization Concept, Exercise and Tape — The technique will be applied to cases in the sham group with only hand contact, without any slippage or rotation in any direction. Then, rigid taping will be applied without any tension or direction, and home exercises will be given.
  Arms: Sham Movement Mobilization Concept Group
Behavioral: Special Exercises — Subjects in the control group will be shown home exercises customized for knee osteoarthritis and asked to continue them.
  Specialized Home Exercises for the Knee Joint
  1. Lumbar extensor stretching, Hamstring stretching, hip flexors stretching, TFL stretching,
  2. Straight leg raise (lying on back and side)
  3. Bridge exercise
  4. Drawing circles while lying on your back and side
  5. Knee flexion-extension
  6. Weight bearing exercises
  7. Tiptoe exercise
  8. Step climbing and descending exercise
  9. Terminal knee extension
  10. Strengthening the muscles around the hips
  Arms: Control Group

SUMMARY:
Individuals with knee osteoarthritis are one of the groups most affected by musculoskeletal disorders and experience pain and mobility limitations that significantly limit their daily living activities. Quantitative sensory assessment in individuals with osteoarthritis plays a critical role in evaluating disease progression and treatment effectiveness by objectively measuring changes in sensory perception such as proprioception and nociception. These changes in sensory perception can negatively affect individuals' movement control and balance. In this context, evaluation of quantitative sensory parameters allows the development of more targeted and effective interventions in the rehabilitation processes of individuals with osteoarthritis.

Additionally, electromyographic evaluation in individuals with osteoarthritis analyzes muscle activation levels, providing a better understanding of the impairments in muscle functions of these individuals. EMG data helps to design rehabilitation programs individually by determining to what degree muscles are activated and which muscle groups are more affected. Decreased muscle activation or abnormal muscle activation in individuals with osteoarthritis can negatively affect joint stability and mobility. Therefore, EMG evaluations are an objective method to evaluate the effectiveness of treatment strategies aimed at restoration of muscle functions in individuals with osteoarthritis.

The quantitative sensory and EMG evaluations performed in this project aim to improve the quality of life of individuals by offering innovative approaches in the clinical management of individuals with osteoarthritis. Therefore, these evaluations are of critical importance for the original value and scientific contribution of our project. For these reasons, the selection of individuals with osteoarthritis and the detailed evaluations made on these individuals and its connection with the methods can be considered as the innovative and original aspect of our project.

The aim of this study is to investigate the effect of the Mulligan movement mobilization concept on quantitative sensory parameters, pain and muscle activation levels in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative disease that occurs especially in weight-bearing joints, characterized by a decrease in joint space due to progressive cartilage loss, subchondral sclerosis and osteophyte formations (Martel et al., 2016). Although OA is also seen in the hip, spine and hand joints, it is most commonly seen in the knee joint (Neogi et al., 2012). Although the primary change in knee OA is in the articular cartilage of the knee, all tissues in and around the joint are affected by OA. The clinical features of the condition are pain, joint stiffness, edema, local tenderness in the joint, crepitation and swelling, muscle weaknesses, osteophytes, instability, subluxations, joint deformities, limitation of joint movement and functional limitations (Sharma 2021).

Pain in knee osteoarthritis is a multifactorial phenomenon in which structural, neurophysiological and psychosocial factors play a role (Emmert et al, 2018). Regarding neurophysiological factors, it has been shown that there are inflammatory mediators within the articular cartilage that alter afferent sensory inputs and cause plastic changes in the nervous system leading to central sensitization (Schaible et al, 2022). Although it is such a multifactorial symptom, the methods used in the evaluation of pain sensation for osteoarthritis are mostly subjective and include the patient's feedback, such as visual analog scale, numerical rating scale, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Knee Injury and Osteoarthritis Outcome Score (KOOS). ) is limited to tests, surveys or scales (Dainese et al, 2022). Although these scales are an important part of clinical practice and reflect the patient's capacity to express his or her own experience, they provide subjective information on issues such as the patient's pain intensity, the effects of pain, and its effects on quality of life (Dainese et al, 2022).

Quantitative sensory testing (QST) is a systematic psychophysical testing method used to measure sensory thresholds for pain, touch, vibration and temperature sensations (Mücke et al, 2021). It measures individual sensory perceptions using direct patient feedback. It tests sensory loss (hypoesthesia, hypoalgesia) and sensory gain (hyperesthesia, hyperalgesia, allodynia) and is used to test the nociceptive and non-nociceptive properties of different afferent nerve fibers and central pathways (Mücke et al, 2021). Quantitative sensory testing may offer a more objective approach to identifying underlying causes of pain. Physical measurements such as nerve damage, loss of sensation, and changes in touch sensitivity can provide more objective data in assessing pain (Arant et al, 2021).

It has been reported that pain, movement limitations and muscle weakness in individuals with osteoarthritis cause indirect effects on muscle activity and functions (Petterson et al, 2023). Changes in muscle activity usually occur in response to pain or as the patient tries to compensate for functional limitations in the joint (Petterson et al, 2023).

It has been shown that due to pain and movement limitations in the affected joint, it causes the individual to change body position and use other muscle groups more (Sharma 2021). Avoidance of using the affected joint has also been reported as a factor in the weakening of the relevant muscle groups. OA can affect joint stability, which can impair muscle coordination (Sharma 2021). Superficial Electromyography (EMG) appears as a method that helps us monitor changes in the activation patterns of certain muscle groups and understand the underlying causes of these functional limitations (Simonsen et al., 2014).

OA treatment generally focuses on relieving symptoms, controlling pain, improving joint function, and improving quality of life (Block et al, 2020). Treatment methods used in the rehabilitation of patients with OA include exercise, electrotherapy and manual therapy. Mulligan Movement Mobilization (MWM), which is among manual therapy practices, is a manual therapy concept developed by Brian Mulligan. This concept includes a set of techniques aimed at correcting pain and limitations in joint range of motion (Anwer et al, 2018). It has been supported by studies that in conditions such as osteoarthritis, these mobilization techniques can help increase joint mobility and relieve the patient's symptoms (Alkhawajah et al, 2019).

The basic principles of Mulligan Movement Mobilization include collaboration with the patient, pain-free mobilization, and a manual force applied during a specific joint movement. It is aimed to increase joint range of motion, pain control and functional recovery, and to contribute to the patient being more effective in daily activities by increasing joint function (Oskay et al., 2015), (Alkhawajah et al., 2019).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosing knee OA according to the American College of Rheumatology (ACR) criteria (Primary knee OA diagnosis)
* Stage 2 or 3 patients according to Kellgren-Lawrence radiological staging criteria
* Patients with a disease duration of 6 months or longer
* Participants aged between 50 and 70
* Being able to walk without using assistive devices
* Body mass index is below 35 kg/m²
* Pain intensity must be between 3 and 7 according to the Numerical Pain Rating Scale
* Not having received physiotherapy in the last year.

Exclusion Criteria:

* Infiltration with steroids or local anesthetics in the year before the patient entered the study or during follow-up
* Obtaining the indication for surgery
* Severe hearing, vision and speech impairment
* Having serious systemic and cardiovascular diseases that prevent exercise
* Having a neurological disease
* Having a lower extremity deformity (severe varus or valgus deformity, significant joint instability and other orthopedic problems requiring surgical intervention)
* Patients with acute knee inflammation
* Having any disorder, syndrome or disease that may cause myofascial or neuropathic pain in the lower extremities, such as lumbar radiculopathy, meralgia paresthetica or Saphenous nerve compression.
* Cognitive deficit (Alzheimer's, dementia) revealed in the clinical history.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of muscle activation: | 2 mounth
  Evaluation of muscle activation with EMG: It will be evaluated with the Noraxon MyoMuscle system. (Noraxon Inc., Scottsdale, AZ, USA) sEMG (Noraxon myosystem DTS, USA) will be used to measure the electrical activity of the muscles. sEMG data of the muscles will be recorded and muscle activities will be analyzed. Ag/AgC superficial electrodes will be used for sEMG measurements. Superficial 8-channel EMG (Bilateral Quadrieps Femoris (rectus femoris, vastus lateralis, vastus medialis), Biceps femoris (long and short head), Semitendinosus).
Pain Sensation and Sensory Evaluation | 2 mounth
  Pressure pain thresholds (BAEs) are measured using a calibrated digital algometer (Algomed/MEDOC) by slowly increasing mechanical pressure at a computer-controlled rate of 1 kg/s.
  To elicit temporal summation in all of the above-mentioned regions, mechanical stimulation was applied 10 times using a digital algometer calibrated at 110% of the pressure pain threshold intensity with a 1-second interstimulus interval. When creating temporal summation, the procedure was started at least 2 minutes after the last PPT was measured to ensure that the tests were not contaminated. Before the first stimulus, study participants were asked to verbally indicate their pain levels at the first, fifth and tenth stimuli according to a visual analogue scale (VAS) placed in front of them. VAS is fixed with single digit numbers from 0 to 10, 0 being "no pain", 1-2 "very mild pain", 3-4 "mild pain", 5-6 "moderate pain", 7-8 " "severe pain" and 9-10 as "very severe unbearable pain".

SECONDARY OUTCOMES:
Muscle strength assessment | 2 mounth
  Muscle strength assessment and maximum voluntary contraction measurement: with Hand Held Dynamometer Quadriceps and Hamistring muscle strength will be measured with a portable manual muscle strength measuring device (Model 01165, Lafayette, IN, USA). (Layefette Instrument®, Layafette,IN).
sit and reach test battery | 2 mounth
  General flexibility of lower extremity muscles: sit and reach test battery
  Sit-Reach Test for Flexibility: The participant was asked to sit with his knees straight, without shoes, and to reach as far forward as he could with his arms and palms facing down, without bending his knees. The distance the participant crosses their toes is measured. The test is repeated 3 times and the best result is recorded in cm (Lemmink et al., 2003).
Timed get up and go test | 2 mounth
  Patients are instructed to sit upright on a standard stool of approximately 45 cm with their feet flat on the floor. With the 'Start' command, patients are told to get up without holding on, walk towards the object 3 meters away, turn around and sit down again. The entire duration is recorded with a stopwatch (Piva et al., 2004).
WOMAC | 2 mounth
  The Western Ontario and McMaster University Arthritis Index (WOMAC) is a patient-reported outcome index for the evaluation of lower extremity OA. The WOMAC index has been used for decades. It is one of the most frequently used outcome measures in research on hip and knee OA. WOMAC has been suggested as one of the highest performing outcome measures for knee and hip OA in terms of reliability, validity, responsiveness, and interpretability (Tüzün et al., 2005).
Tampa kinesiophobia scale | 2 mounth
  Chronic pain may cause behavioral changes due to physical and psychological reasons. The Tampa Kinesiophobia Scale score range is 17 to 68, with a higher score indicating increased kinesiophobia. The psychometric properties of the Tampa Kinesiophobia Scale have been tested in many different languages and have been used for many different musculoskeletal pains (Yılmaz et al., 2011).

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No